CLINICAL TRIAL: NCT07331766
Title: Effectiveness of a Novel Cross Sectorial Collaborative Treatment Pathway for Chronic Pain Patients. A Multicenter Randomized Controlled Trial.
Brief Title: Collaboratory Treatment Pathway for Chronic Pain Patients.
Acronym: PainPath
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital of North Norway (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Astrid Woodhouse, Associate Professor, St. Olavs Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 898717; 024201 (Other Grant/Funding Number: Klinbeforsk, Norway)
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Chronic (Non-malignant) Musculoskeletal Pain; Patients Referred to Multidisciplinary Pain Clinics
Keywords: chronic pain; multidisciplinary pain clinic; Standardized treatment pathway; collaboration across levels of health care; collaboration
MeSH Terms: conditions — Chronic Pain; Bronchiolitis Obliterans Syndrome; Musculoskeletal Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A collaborative treatment pathway for patients referred to multidisciplinary pain clinics. (Experimental): The study intervention is a new standardized treatment pathway with exteded collaboration for patients referred to pain clinics.
  Interventions: Other: A collaborative treatment pathway for patients referred to multidisciplinary pain clinics in Norway
- Treatment as usual: Standard care at a multidisciplinary pain clinic (Active Comparator): Standard care following present procedures at the multidisciplinary pain clinics involved in this study
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: A collaborative treatment pathway for patients referred to multidisciplinary pain clinics in Norway — The study intervention is a standardized treatment pathway for patients referred to multidisciplinary pain clinics. The pathway is designed to support structured collaboration across health care levels and other sectors. It includes two digital multidisciplinary meetings with the patient, the pain clinic, and additional stakeholders, such as social security representatives. The pathway delineates a clearly defined course of treatment with scheduled follow-up over a six-month period.
  Arms: A collaborative treatment pathway for patients referred to multidisciplinary pain clinics.
Other: Treatment as usual — The comparator intervention reflects the current standard of care provided at four Norwegian pain clinics. Standard care may vary slightly between clinics but generally includes a multidisciplinary clinical evaluation involving at least two different healthcare professions. A clinical summary outlining recommendations for further follow-up is sent to the referring physician. Most patients also receive a summary consultation with the pain clinic team, and some are offered additional treatment at the pain clinic.
  Arms: Treatment as usual: Standard care at a multidisciplinary pain clinic

SUMMARY:
In this multicenter randomized controlled trial, the aim is to evaluate the effectiveness of a standardized treatment pathway (STP) for patients referred to four participating pain clinics, by comparing it to treatment as usual (TAU) which is standard care at the clinics.

The STP differs from TAU in two key aspects:

* Structured cross-sector collaboration: Involvement of primary healthcare providers, particularly the patient's GP, in two digital collaborative meetings with the pain clinic.
* Time-bound treatment pathway: A clearly defined treatment trajectory with follow-up over a six-month period.

The study aims to answer whether the STP give larger improvements than TAU in the following outcomes:

* patients´ reported overall impression of change in health (primary outcome)
* pain interference (primary outcome)
* physical function and mental health
* satisfaction with and experience of continuity and integration of the health care services

All study participants will follow an initial care pathway at the pain clinic, which includes:

* a screening consultation with a study coordinator
* a multidisciplinary clinical assessment based on a biopsychosocial approach by at least to health care professions. The specific professional groups included in each assessment are determined individually based on patient needs.

The control group:

This group will receive standard care at the pain clinic. This will vary somewhat between the four pain clinics , but almost all patients will be offered a summary consultation with the pain clinic team where further plans for follow-up will be discussed. Some patients will be offered further treatment at the pain clinic.

All clinics will send a clinical summary to the referring physician with suggestions for further follow-up. If further collaboration with primary care is needed, it may preferably be written or arranged via telephone. Digital collaborative meeting will not be offered to this group.

The intervention group:

All patients in this group will be offered the STP with two digital collaborative meetings as described above.

DETAILED DESCRIPTION:
A new standardized treatment pathway (STP) has been developed by the Pain Research Group at St. Olav's Hospital. The STP is designed to establish structured collaboration between specialist and municipal health services, as well as the Norwegian Labor and Welfare Administration (Nav). In this study, the STP will be compared to the current standard of care, which typically involves multidisciplinary clinical assessments followed by a summary consultation between the pain clinic and the patient.

The key innovation of the STP lies in its cross-sectorial collaboration, most notably the inclusion of the patient's general practitioner (GP) in two structured video consultations with the patient and the multidisciplinary pain clinic. When relevant, a Nav representative or representatives from municipal and specialized health service may also participate. A collaborative treatment plan is developed during the first video consultation and reinforced through a six-month follow-up period, culminating in a second collaborative consultation.

Given that the STP is more resource-demanding than current practices at Norwegian pain clinics, involving coordinated efforts across multiple sectors, it is crucial to evaluate its overall effectiveness. Equally important is identifying which patient subgroups may benefit most from this approach, to ensure that resources are allocated efficiently and care is tailored to those with the greatest need.

The primary aim of this study is to evaluate the effectiveness of the STP for patients referred to one of four participating pain clinics, by comparing it to TAU in a randomized controlled trial.

Hypotheses, aims and objectives:

The primary aim of this study is to investigate if patients with chronic pain admitted to a pain clinic and who receive a new collaborative STP will have larger improvements in overall impression of change in health and pain interference compared to patients who receive TAU.

Hypotheses: Compared to the control group, we hypothesize that patients in the intervention group will report:

H1) less pain interference H2) better overall change in health

The secondary aims of the study are to compare collaborative STP with TAU in terms of:

Aim 1: physical functioning Aim 2: mental health Aim 3: participants' experience of continuity and integration of the health care services Aim 4: participants' satisfaction with the health care services and social security services Aim 5: prescriptions of opioids and other potentially addictive medication Aim 6: use of primary and specialist health care Aim 7: return to work and decisions from Nav Aim 8: referring GPs' satisfaction with the pain clinic management

Hypotheses (for secondary aims): Patients in the intervention group will have/report:

* better physical functioning and mental health (aim 1, 2)
* better experiences of continuity and integration of health care services (aim 3)
* more trust in health care services and social security services (aim 3)
* better collaboration between health care services and social security services (aim 3)
* higher overall satisfaction with the GP, the pain clinic treatment and social security services (aim 4)
* higher probability of reducing the use of opioids and other potentially addictive medications (aim 5)
* differences in consultation frequency in specialist health care and primary health care (aim 6)
* higher probability of (re)entry to competitive work or education (and fewer days on sick leave / working allowance / benefits / disability / pension), when applicable, and a shorter time to being granted disability pension, when applicable (aim 7)
* The GPs of patients in the intervention group will report higher satisfaction with the pain clinic management (aim 8)

Project methodology:

This is a multi-center study that will include patients with chronic and complex pain undergoing treatment at one of four multidisciplinary pain clinics in Norway: St. Olav's hospital, Haukeland University hospital, University hospital in Northern Norway and Innlandet Hospital.

Design:

The study is a two-group randomized controlled study comparing a new collaborative STP with usual care at four multidisciplinary pain clinics. Each clinic will randomize their patients into an intervention group (collaborative STP) and a control group (TAU).

Study sample:

A total of 386 patients will be included in the study (see sample size estimation).

Inclusion criteria:

Patients aged 18-80 years with an accepted referral for multidisciplinary care by one of the four pain clinics.

Exclusion criteria:

Patients referred for monodisciplinary care are not eligible for this study. Participants who are unable to perform the required tasks or procedures necessary for participation in the study will be excluded. These tasks include, but are not limited to, completing questionnaires that, due to technical reasons, are available only in Norwegian language, and being capable of participating meaningfully in collaborative meetings as assessed by clinical professionals.

Additionally, patients who have already undergone a mapping consultation (see next section) and have been deemed ineligible for further follow-up at the pain clinic will also be excluded from participation.

Inclusion, informed consent and randomisation:

Initial information:

All patients who meet the admission criteria for multidisciplinary care at the pain clinic will receive a general admission letter with information about the clinic and the scheduled times for clinical consultations. Patients who are eligible for the study will receive a separate letter containing written information about the study.

In order to find eligible patients, we applied to the Regional Committee for Medical and Health Research Ethics (REK) and the study was given an exemption from the duty of confidentiality. This exemption will allow digital distribution of study information to patients, based on data extracted from their medical records.

All personal data related to individuals who do not consent to participate, do not attend the screening consultation, or do not respond to the invitation within three weeks will be deleted continuously and without delay.

The study information package will include:

1. the scheduled time for a screening consultation with the local study coordinator, where further information will be provided and eligibility for study inclusion will be assessed
2. a study information letter, including details on data handling in accordance with GDPR and national regulations
3. a consent form
4. notification of an upcoming phone call from the study coordinator, inviting the patient to the screening consultation

This information will be sent digitally via the secure platforms "helsenorge.no" or "HelsaMi"

Patients will be given the following options:

1. decline participation based on the written information
2. await the phone call from the study coordinator and either accept or decline participation based on the information provided
3. attend the screening consultation before making a decision
4. ignore the phone call and the screening consultation, thereby opting out of inclusion

In some cases, the clinic may require additional information before confirming eligibility for care. These patients will be scheduled for a digital screening consultation with a clinician. Only those admitted to further contact with the clinic will proceed to the screening consultation.

The study coordinator's screening consultation:

Before the first clinical consultation, eligible patients will be contacted by a study coordinator via telephone and invited to a screening consultation, scheduled at least one week after the initial information package to allow time for consideration.

During the coordinator's screening consultation:

* The study information will be repeated orally
* Patients will have the opportunity to ask questions
* Written informed consent will be obtained if they choose to participate
* Participants will receive contact information for the study coordinator and be reminded that participation is voluntary and can be withdrawn at any time without consequences for their care at the pain clinic

Finally, participants will be randomized using the digital randomization system provided by eFORSK. The randomization will be stratified according to clinic. A block randomization method with permuted blocks of random sizes (e.g. 4 to 8 subjects) will be used. The allocation ratio between the intervention and control groups will be 1:1.

The intervention and the control group:

All study participants will follow an initial care pathway at the pain clinic, which includes:

* a screening consultation (if necessary)
* the screening consultation with a study coordinator
* a multidisciplinary clinical assessment based on a biopsychosocial approach. In this study, multidisciplinary is defined as involving two or more clinical professions. The specific professional groups included in each assessment are determined individually based on patient needs.

The control group

Participants in the control group receive standard care at the pain clinic, which includes:

* a multidisciplinary clinical evaluation involving at least two different clinical professions
* a clinical summary sent to the referring physician
* a summary consultation between the patient and the multidisciplinary team at the pain clinic is offered to most of the participants (not obligatory at one of the pain clinics).

Primary care representatives do not participate in the summary consultation for the control group. A clinical summary is sent to the referring physician (most commonly patient's general practitioner) detailing either the planned treatment at the pain clinic or recommendations for further follow-up in municipal health services or other specialist healthcare services. If further collaboration with primary care is needed, it may preferably be written or arranged via telephone.

The intervention group: Standardised Treatment Pathway (STP) Participants in the intervention group receive a similar initial care pathway as the control group, including the screening consultation and multidisciplinary clinical evaluation, in accordance with the National Pathway for Chronic and Complex Pain Conditions.

The intervention consists of three steps:

Patients and their GPs will be informed as soon as they are randomized to the intervention group about the intervention. This will be done by a separate information sheet to the patients, and a letter with general information to the GP about the study and suggested time and date for the first collaborative consultation. Following this, the intervention group gets the multidisciplinary clinical assessment and engages in a pre-planned digital collaborative consultation arranged by the pain clinic. This consultation includes:

* the patient's GP, and when relevant:
* representatives from municipal and specialised health services
* the patient's Nav coordinator The patient can also choose to invite a relative to participate in this consultation.

During the consultation, a comprehensive treatment plan is developed collaboratively, covering a six-month follow-up period. This plan may include:

* consultations with the GP
* local physiotherapist or other primary health care services
* follow-up by Nav, the pain clinic, or other specialist healthcare providers The care pathway concludes with a second collaborative consultation approximately six months later. This meeting includes the patient, their GP, and one or more of the same health care providers from the pain clinic. Other stakeholders involved in the treatment may also be invited to participate. The purpose of this final consultation is to evaluate progress and adjust the treatment plan if needed.

Statistical analyses The primary analysis will estimate difference in either means or proportions with 95% confidence interval (CI) between the intervention and control groups over the first 6 and 18 months. The analyses will be conducted according to the intention to treat principle using a linear mixed model for differences in means and generalised estimating equations (GEE) for differences in proportions. In the mixed models, correlation between repeated observations within individuals and correlation between patients having the same GP are accounted for by specifying random effects.

The effect of the intervention and time will be specified as fixed effect using a joint variable of intervention and time. Here, baseline levels are pooled over the two study groups assuming that any baseline differences are due to chance. In the GEE models, correlations between repeated observations between individuals are accounted for by specifying a correlation structure. The effect will be estimated both crude and adjusted for study center, which will be used to stratify the randomisation, as well as other important prognostic factors (e.g., age, sex, educational level and clinical characteristics).

Missing values are inherently accounted for in the GEE and mixed model approach by including all available information, but multiple imputation methods and complete case analysis will be applied in sensitivity analyses. Additional protocol analysis will be specified in the statistical analysis plan for the trial. The decision on which variable to inform on adherence is guided by experience from the feasibility study. Stratified analyses of the primary outcome will be performed as secondary analyses. Analyses may include stratification for gender, age-groups, socioeconomic status, etc.

Most secondary outcomes will be analysed using a similar approach as described for the primary outcome with linear mixed models. Time to sustainable return to work will be analysed using Cox regression.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older who have been granted the right to specialist health care in accordance with the Norwegian National prioritization guideline for pain clinics, and who are scheduled for multidisciplinary treatment involving at least two professionals from the pain clinic.

Exclusion Criteria:

Patients scheduled for monodisciplinary treatment. Patients referred solely for invasive procedures. Patients without sufficient language skills to understand the study information and provide informed consent. Patients are excluded if interpreter services are required.

Patients deemed unable to complete study-related tasks (e.g., questionnaires). Patients referred exclusively for stabilization or tapering of opioids or other medications considered addictive.

Patients who will be unable to participate in collaborative meetings or follow the treatment plan due to extensive ongoing or planned care trajectories within other specialist health services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain interference | At baseline and through to 18 months after baseline
  Pain interference questions (q8-q14)from the Brief Pain Inventory questionnaire (BPI)
Overall impression of change in health | Measured 18 months after baseline
  Patient global impression of change questionnaire (PGIC)

SECONDARY OUTCOMES:
Physical function | From baseline and to 18 months after baseline
  Physical function domain from the PROMIS-29 questionnaire and Oswestry disability questionnaire (generic version)
Mental health | From baseline to 18 months after baseline
  Mental health domain from the PROMIS-29 questionnaire
Patient experience of continuity and integration of health care services | From baseline to 18 months after baseline
  The IntegRATE questionnaire, 4 items
Trust in health care services and social security services | From baseline to 18 months after baseline
  In-house questions on patients' trust in the services
Collaboration between health care services | From baseline to 18 months after baseline
  In-house question on patients' experiences about the GP's collaboration with others
Satisfaction with the patient's GPs | From baseline to 18 months after baseline
  Five in-house questions on the patients satisfaction with GP. 3 items
Patient's satisfaction with the pain clinic | From 2 weeks after 1.st collaborative meeting/ summary meeting to 18 months after baseline
  In-house question on patient satisfaction. 1 item
Use of prescibed opioids or other potentially addictive medications | From baseline to 18 months after baseline
  Data will be collected from a national registry over prescribed medication
Health care utilisation, specialist health care | From baseline to 18 months after baseline
  Registry data: Number of outpatient visits, number of days with day treatment, number of in-patient days.
Health care utilisation, primary health care | From baseline to 18 months after baseline
  Registry data: Number of GP ordinary consultations, number of other GP contacts, number of out-of hour visits
Return to work and other decisions from the Norwegian social security systems (Nav) | from baseline to 18 months after baseline.
  Registry data on (re)entry to competitive work or education; days on sickleave; working allowance benefits; disability pension, time frame for decisions
Sleep problems | From baseline to 18 months after baseline
  The sleep domain from PROMIS29
Pain intensity | From baseline to 18 months after baseline
  Pain intensity the past week: strongest pain, weakest pain, mean pain and pain right now. First five questions from the Brief Pain Inventory.

OTHER OUTCOMES:
The referring GP's satisfaction with the pain clinic management | From within 2 weeks after summary consultation (control group)/ collaborative consultation (intervention group) to 12 months after baseline
  In-house questionnaire to GP
Pain locations | From baseline to 18 months after baseline
  Body locations with pain: a check list from the NorPain registry (a national quality registry for pain clinics)
Severity of symptoms of fatigue, depression, memory/concentration, sleep problems, headache and stomach pain | From baseline to 18 months after baseline
  The questions are from the Symptom severity scale - in use for the classification of Fibromyalgia syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Woodhouse, Phd, Principal Investigator — St Olavs Hospital/ Smertesenteret; Mari Glette, PhD, Study Chair — St. Olavs Hospital; Tormod Landmark, PhD, Study Chair — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Innlandet Hospital, Ottestad, Innlandet
  - University Hospital of Northern Norway, Tromsø, Troms
  - St Olavs hospital, Trondheim, Trøndelag
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the approved informed consent does not permit data sharing beyond the study team, and applicable data protection regulations (including GDPR) restrict secondary transfer of participant-level health data without explicit consent.

REFERENCES:
- See also: The published version of the National treatment path for patients referred to multidisciplinary pain clinics in Norway — https://www.helsedirektoratet.no/nasjonale-forlop/smerte
- See also: Project information site (in Norwegian language). This site is shared with GP's when invited to participate in collaborative meetings. — https://www.smertenettverk.no/painpath